CLINICAL TRIAL: NCT01713959
Title: Feasibility Study: Evaluation of the Safety and Efficacy of the Ulthera® System for the Treatment of Axillary Hyperhidrosis
Brief Title: Feasibility Study: Ulthera® System for the Treatment of Axillary Hyperhidrosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ulthera, Inc (Industry)
Responsible Party: Sponsor
Organization: Merz North America, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ULT-121
Record Dates: First submitted 2012-10-15; First posted 2012-10-25 (Estimated); Last update posted 2017-11-24 (Actual); Status verified 2013-06

CONDITIONS: Hyperhidrosis
Keywords: Underarm sweating
MeSH Terms: conditions — Hyperhidrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A - Split Body Treatment (Experimental): Active treatment of one axilla with the Ulthera System Treatment; Sham treatment of one axilla.
  Interventions: Device: Ulthera System treatment; Device: Sham treatment
- Group B: Ulthera System Treatment w lido (Active Comparator): Subjects receive a bilateral Ulthera System Treatment, with one axilla receiving a subcutaneous lidocaine injection.
  Interventions: Device: Ulthera System treatment

INTERVENTIONS:
Device: Ulthera System treatment — Ulthera System: Focused ultrasound energy delivered below the surface of the skin.
  Other Names: Ulthera® System; Ultherapy™ Treatment; Ulthera, Inc.; Ultrasound treatment for skin tightening
Device: Sham treatment — Sham Treatment: Use of the Ulthera System with the system adjusted to deliver 0 energy.
  Arms: Group A - Split Body Treatment

SUMMARY:
Single-center, randomized, split-body, pilot study, treatment of up to 23 subjects in two treatment groups. Subjects will receive two Ultherapy treatments at Day 0 with follow-ups at 7 and 14 days post-treatment #1, and Day 28 with follow-ups are 7, 14, 30, 60, 90 days post-treatment #2.

DETAILED DESCRIPTION:
Subjects will be randomized to one of two study groups:

* Group A: Split body treatment. Ultherapy to one axilla, Sham treatment to the other axilla.
* Group B: Bilateral Ultherapy treatments, with a pre-treatment subcutaneous lidocaine injection administered to one axillary side.

Hyperhidrosis Disease Severity Scale (HDSS), gravimetric test and starch iodine test will be obtained at all study visits. Patient satisfaction questionnaires will also be obtained at 30, 60 and 90 days post-treatment #2.

ELIGIBILITY:
Inclusion Criteria:

* Male and female, ages 18-75
* Subject is in good health
* Diagnosis of bilateral axillary hyperhidrosis refractory to previous topical therapies
* At least 50 mg of spontaneous resting axillary sweat production in each axilla measured gravimetrically at room temperature/humidity (20 - 25.6°C/20-80%) over a period of 5 minutes. (Patients should be at rest for at least 30 minutes after physical exercise including walking.)
* HDSS score of 3 or 4.
* Understands and accepts the obligation not to undergo any other procedures in the areas to be treated through the follow-up period.

Exclusion Criteria:

* Dermal disorder including infection at anticipated treatment sites in either axilla.
* Previous botulinum toxin treatment of the axilla in the past year.
* Expected use of botulinum toxin for the treatment of any other disease during the study period.
* Known allergy to starch powder or iodine.
* Secondary hyperhidrosis, for example, hyperhidrosis that is secondary to other underlying diseases including hyperthyroidism, lymphoma and malaria.
* Previous surgical treatment of hyperhidrosis including sympathectomy, surgical debulking of the sweat glands, subcutaneous tissue curettage and ultrasonic surgery.
* Women who are pregnant, lactating, possibly pregnant or planning a pregnancy during the study period.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2011-08; Primary Completion 2012-04 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Improvement in sweat production | 90-days post-treatment treatment #2
  Axillary hyperhidrosis as assessed by using a gravimetric method.

SECONDARY OUTCOMES:
Improvement in sweat production at follow-up timepoints other than 90 days post-treatment | Participants will be followed up to 60 days post-treatment
  Axillary hyperhidrosis as assessed by using a gravimetric method.
Area of efficacy | Participants will be followed for up to 90 days following treatment #2.
  Starch iodine test will be used to assess the area of efficacy. Imaging will be obtained.
Qualitative measure of hyperhidrosis severity | Participants will be followed for up to 90 days following treatment #2
  The HDSS is a scale used for primary axillary/underarm hyperhidrosis patients. It provides a qualitative measure of the severity of their condition based on how it affects their daily activities. Patients select the statement that best reflects their experience with underarm sweating.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Nestor, MD, Ph.D, Principal Investigator — The Center for Clinical & Cosmetic Research
Locations (1):
- The Center for Clinical & Cosmetic Research, Aventura, Florida, United States